CLINICAL TRIAL: NCT01286558
Title: An Eight-week Randomised Double-blind Study to Compare the Efficacy and Safety of Telmisartan 80mg Plus Amlodipine 5 mg Fixed-dose Combination vs. Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination in Patients With Hypertension
Brief Title: Comparison in Japan T80/A5 (Telmisartan 80 mg and Amlodipine 5 mg) and T40/A5 (Telmisartan 40 mg and Amlodipine 5 mg)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1235.37
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine

ARMS (2):
- 80mg telmisartan and 5mg amlodipine FDC (Experimental): once daily
  Interventions: Drug: 5 mg amlodipine; Drug: 80 mg telmisartan
- 40mg telmisartan and 5mg amlodipine FDC (Active Comparator): once daily
  Interventions: Drug: 40 mg telmisartan; Drug: 5 mg amlodipine

INTERVENTIONS:
Drug: 40 mg telmisartan — once daily
  Arms: 40mg telmisartan and 5mg amlodipine FDC
Drug: 5 mg amlodipine — once daily
  Arms: 80mg telmisartan and 5mg amlodipine FDC
Drug: 5 mg amlodipine — once daily
  Arms: 40mg telmisartan and 5mg amlodipine FDC
Drug: 80 mg telmisartan — once daily
  Arms: 80mg telmisartan and 5mg amlodipine FDC

SUMMARY:
Blood pressure in hypertensive patients is rarely controlled to an optimal level by one drug alone, often a combination of two or more drugs is essential to achieve a sufficient antihypertensive effect. Therefore in Japanese Society of Hypertension (JSH) 2009 combination therapy is recommended. In JSH 2009 it is advised to start the combination therapy at a low dose, and to increase the dosage when the antihypertensive effect is not sufficient. In the Japanese long-term safety study, 259 patients received the T40/A5 mg fixed-dose combination (FDC), and after 6 weeks treatment 48 patients of them could not control their blood pressure (DBP =90) (U09-2494-01). For those patients who cannot control their blood pressure with T40/A5 mg FDC, a switch to a higher dose such as T80/A5 mg is recommended.

In the overseas 4x4 factorial design trial, a clinically meaningful difference of the blood pressure lowering effect between T80/A5 mg free combination and T40/A5 mg free combination was shown (U07-3503-02). But the sponsor has no data that verifies this difference in Japanese patients.

Thus, this clinical trial is being conducted to investigate the antihypertensive effect and safety of high dose T80/A5 mg FDC compared with low dose T40/A5 mg FDC in Japanese patients with essential hypertension. In this trial, a multi-centre, randomised, double-blind, double-dummy, active-controlled, parallel group comparison method is employed.

ELIGIBILITY:
Inclusion criteria:

1. Essential hypertensive patients

   * If already taking antihypertensive drugs, mean seated diastolic blood pressure (DBP) must be >=90 and >=114 mmHg
   * If not taking any antihypertensive drugs, mean seated DBP must be >=95 and >=114 mmHg
2. Able to stop all current antihypertensive drugs without risk to the patient based on the investigators opinion.

Exclusion criteria:

1. Patients taking 3 or more antihypertensive drugs at signing the informed consent form
2. Patients with known or suspected secondary hypertension
3. Patients with clinically relevant cardiac arrhythmia
4. Congestive heart failure with New York Heart Association (NYHA) functional class III-IV
5. Patients with recent cardiovascular events
6. Patients with a history of stroke or transient ischaemic attack within last 6 months before signing the informed consent form
7. Patients with a history of sudden deterioration of renal function with angiotensin II receptor blockers (ARBs) or angiotensin converting enzyme (ACE) inhibitors; or patients with post-renal transplant or post-nephrectomy
8. Patients who have previously experienced characteristic symptoms of angioedema (such as facial, tongue, pharyngeal, or laryngeal swelling with dyspnea) during treatment with ARBs or ACE inhibitors
9. Patients with known hypersensitivity to any component of the investigational product, or a known hypersensitivity to dihydropyridine-derived drugs
10. Patients with hepatic and/or renal dysfunction
11. Pre-menopausal women who are nursing or pregnant

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (8):
- Japan (8):
  - 1235.37.01 Boehringer Ingelheim Investigational Site, Chuo-ku,Tokyo
  - 1235.37.07 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 1235.37.08 Boehringer Ingelheim Investigational Site, Itoshima, Fukuoka
  - 1235.37.02 Boehringer Ingelheim Investigational Site, Katsushika-ku, Tokyo
  - 1235.37.05 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1235.37.03 Boehringer Ingelheim Investigational Site, Ota-ku, Tokyo
  - 1235.37.06 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1235.37.04 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Started | 112 | 113
Completed | 111 | 111
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC | Total
Number analyzed (Participants) | 112 | 113 | 225
Age, Continuous [Mean (Standard Deviation); unit: year] | 54.6 (8.4) | 52.8 (9.4) | 53.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 89 | 89 | 178

OUTCOME MEASURES:

1. Primary Outcome: Reduction From the Reference Baseline in Mean Seated Diastolic Blood Pressure (DBP) at Trough
Description: Reference baseline: Status of patients after the 12-week open-label run-in period with telmisartan monotherapy followed by 40 mg telmisartan and 5 mg amlodipine combination therapy, where patients' eligibility to enter the double-blind treatment period was examined At trough: 24-hour post-dosing
Time Frame: Reference baseline, 8 weeks
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 112 | 112
mm Hg | 4.93 (0.61) | 3.47 (0.61)
Statistical Analysis 1: Comparison: 80 mg Telmisartan and 5 mg Amlodipine FDC vs 40 mg Telmisartan and 5 mg Amlodipine FDC; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 1.46, 95% CI [-0.22 to 3.14]

2. Secondary Outcome: Reduction From the Reference Baseline in Mean Seated Systolic Blood Pressure (SBP) at Trough
Description: as for outcome 1
Time Frame: Reference baseline, 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 112 | 112
mm Hg | 5.55 (0.90) | 3.41 (0.91)
Statistical Analysis 1: Comparison: 80 mg Telmisartan and 5 mg Amlodipine FDC vs 40 mg Telmisartan and 5 mg Amlodipine FDC; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 2.14, 95% CI [-0.36 to 4.64]

3. Secondary Outcome: Changes From the Reference Baseline in the 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Mean (Relative to Dose Time) for DBP
Description: Reference baseline: Status of patients after the 12-week open-label run-in period with telmisartan monotherapy followed by 40 mg telmisartan and 5 mg amlodipine combination therapy, where patients' eligibility to enter the double-blind treatment period was examined
Time Frame: Reference baseline, 8 weeks
Population: ABPM set, i.e., a subset of FAS and with patients who had available ABPM measurements
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 105 | 107
mm Hg | -1.54 (0.49) | -0.33 (0.49)
Statistical Analysis 1: Comparison: 80 mg Telmisartan and 5 mg Amlodipine FDC vs 40 mg Telmisartan and 5 mg Amlodipine FDC; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.21, 95% CI [-2.58 to 0.15]

4. Secondary Outcome: Changes From the Reference Baseline in the 24-hour ABPM Mean (Relative to Dose Time) for SBP
Description: as for outcome 3
Time Frame: Reference baseline, 8 weeks
Population: ABPM set, i.e., a subset of FAS and with patients who had available ABPM measurements
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 105 | 107
mm Hg | -2.81 (0.81) | -0.91 (0.82)
Statistical Analysis 1: Comparison: 80 mg Telmisartan and 5 mg Amlodipine FDC vs 40 mg Telmisartan and 5 mg Amlodipine FDC; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.90, 95% CI [-4.16 to 0.35]

5. Secondary Outcome: Changes From the Pseudo-baseline in the 24-hour ABPM Mean (Relative to Dose Time) for DBP
Description: Pseudo-baseline: Status of patients after the 6-week open-label run-in period with telmisartan monotherapy, where patients' eligibility to enter the double-blind treatment period was examined
Time Frame: Pseudo-baseline, 14 weeks
Population: ABPM set, i.e., a subset of FAS and with patients who had available ABPM measurements
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 105 | 107
mm Hg | -12.16 (0.61) | -11.28 (0.60)
Statistical Analysis 1: Comparison: 80 mg Telmisartan and 5 mg Amlodipine FDC vs 40 mg Telmisartan and 5 mg Amlodipine FDC; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.89, 95% CI [-2.57 to 0.79]

6. Secondary Outcome: Changes From the Pseudo-baseline in the 24-hour ABPM Mean (Relative to Dose Time) for SBP
Description: as for outcome 5
Time Frame: Pseudo-baseline, 14 weeks
Population: ABPM set, i.e., a subset of FAS and with patients who had available ABPM measurements
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 105 | 107
mm Hg | -20.96 (0.96) | -19.32 (0.95)
Statistical Analysis 1: Comparison: 80 mg Telmisartan and 5 mg Amlodipine FDC vs 40 mg Telmisartan and 5 mg Amlodipine FDC; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.64, 95% CI [-4.27 to 0.99]

7. Secondary Outcome: Changes From the Reference Baseline in DBP Hourly Mean Over the 24-hour Dosing Interval as Measured by ABPM
Description: as for outcome 3
Time Frame: Reference baseline, 8 weeks
Population: ABPM set, i.e., a subset of FAS and with patients who had available ABPM measurements
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 105 | 107
mm Hg
  Hour 1 | -1.04 (10.27) | -0.22 (12.38)
  Hour 2 | -1.95 (11.44) | 0.32 (10.93)
  Hour 3 | -2.25 (11.86) | 2.87 (11.61)
  Hour 4 | -3.69 (12.43) | -0.02 (10.63)
  Hour 5 | -1.39 (13.22) | -0.75 (14.06)
  Hour 6 | -1.58 (11.08) | -0.86 (13.32)
  Hour 7 | -0.40 (12.24) | -1.25 (13.22)
  Hour 8 | -1.58 (13.23) | 0.55 (13.83)
  Hour 9 | -2.77 (12.83) | -0.73 (12.44)
  Hour 10 | -2.80 (13.75) | -0.14 (11.58)
  Hour 11 | -1.47 (11.58) | -1.16 (12.05)
  Hour 12 | -0.74 (11.86) | -1.43 (13.65)
  Hour 13 | -2.33 (12.96) | -1.05 (12.03)
  Hour 14 | -0.53 (15.49) | -0.08 (11.36)
  Hour 15 | -0.36 (13.65) | 1.86 (10.88)
  Hour 16 | -0.01 (10.73) | 0.85 (10.97)
  Hour 17 | 0.70 (12.16) | -0.80 (11.07)
  Hour 18 | -1.89 (11.81) | 1.02 (10.33)
  Hour 19 | -3.12 (12.96) | 0.10 (10.38)
  Hour 20 | 0.23 (11.03) | -1.27 (11.93)
  Hour 21 | -3.25 (12.85) | -0.90 (10.81)
  Hour 22 | -2.00 (11.83) | -1.67 (13.14)
  Hour 23 | -2.07 (12.05) | -0.53 (11.95)
  Hour 24 | -0.82 (9.37) | 0.42 (11.23)

8. Secondary Outcome: Changes From the Reference Baseline in SBP Hourly Mean Over the 24-hour Dosing Interval as Measured by ABPM
Description: as for outcome 3
Time Frame: Reference baseline, 8 weeks
Population: ABPM set, i.e., a subset of FAS and with patients who had available ABPM measurements
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 105 | 107
mm Hg
  Hour 1 | -6.54 (16.03) | -1.78 (16.37)
  Hour 2 | -2.78 (14.98) | -0.28 (15.82)
  Hour 3 | -3.41 (16.83) | 2.72 (17.74)
  Hour 4 | -4.72 (18.42) | -1.88 (17.03)
  Hour 5 | -1.14 (18.23) | -2.54 (20.71)
  Hour 6 | -1.68 (18.39) | -2.48 (20.01)
  Hour 7 | -0.60 (19.12) | -2.45 (18.69)
  Hour 8 | -2.05 (20.40) | -0.27 (22.07)
  Hour 9 | -3.09 (17.35) | -1.17 (18.33)
  Hour 10 | -5.78 (19.61) | -0.70 (18.91)
  Hour 11 | -2.04 (19.59) | 0.69 (15.16)
  Hour 12 | -4.57 (17.54) | 0.61 (16.89)
  Hour 13 | -2.27 (19.90) | 0.26 (17.53)
  Hour 14 | -1.46 (21.12) | -1.09 (17.49)
  Hour 15 | -1.21 (17.86) | 1.41 (17.70)
  Hour 16 | -0.78 (17.18) | 0.68 (15.42)
  Hour 17 | -0.71 (17.58) | -1.16 (15.67)
  Hour 18 | -2.66 (18.90) | 1.01 (15.84)
  Hour 19 | -4.58 (18.92) | -1.24 (15.30)
  Hour 20 | 0.57 (19.07) | -3.56 (17.02)
  Hour 21 | -4.02 (17.27) | -1.20 (16.47)
  Hour 22 | -3.88 (16.81) | -4.12 (17.40)
  Hour 23 | -4.65 (21.01) | -2.71 (16.15)
  Hour 24 | -2.24 (16.51) | 0.29 (16.09)

9. Secondary Outcome: Seated DBP Control Rate at Trough
Description: DBP control rate: The rate of patients with controlled seated DBP at trough of less than 90 mmHg after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: Patients included in FAS and with seated DBP >=90 mmHg at reference baseline
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 49 | 50
percentage of participants
  No | 53.1 | 60.0
  Yes | 46.9 | 40.0

10. Secondary Outcome: Seated SBP Control Rate at Trough
Description: SBP control rate: The rate of patients with controlled seated DBP at trough of less than 140 mmHg after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: Patients included in FAS and with seated SBP >=140 mmHg at reference baseline
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 29 | 38
percentage of participants
  No | 55.2 | 55.3
  Yes | 44.8 | 44.7

11. Secondary Outcome: Seated DBP Response Rate at Trough
Description: DBP response rate: The rate of patients who achieved an adequate response in seated DBP at trough (<90 mmHg and/or reduction from reference baseline >=10 mmHg) after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 112 | 112
percentage of participants
  No | 29.5 | 32.1
  Yes | 70.5 | 67.9

12. Secondary Outcome: Seated SBP Response Rate at Trough
Description: SBP response rate: The rate of patients who achieved an adequate response in seated SBP at trough (<140 mmHg and/or reduction from reference baseline >=20 mmHg) after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 112 | 112
percentage of participants
  No | 19.6 | 17.9
  Yes | 80.4 | 82.1

13. Secondary Outcome: Seated Blood Pressure (BP) Normalisation at Trough
Description: Seated blood pressure (BP) normalisation: The numbers of patients whose blood pressure was within normalisation criterion in terms of seated blood pressure after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Number analyzed (Participants) | 112 | 112
participants
  No | 41 | 44
  Optimal | 21 | 13
  Normal | 23 | 26
  High-normal | 27 | 29

ADVERSE EVENTS:
Time Frame: From first drug administration in the double-blind treatment period until 24 hours after the last dose, up to 69 days
Arm/Group | 80 mg Telmisartan and 5 mg Amlodipine FDC | 40 mg Telmisartan and 5 mg Amlodipine FDC
Serious Adverse Events (participants affected / at risk) | 1/112 | 1/113
Other Adverse Events (participants affected / at risk) | 6/112 | 6/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 80 mg Telmisartan and 5 mg Amlodipine FDC (N=112) | 40 mg Telmisartan and 5 mg Amlodipine FDC (N=113)
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 80 mg Telmisartan and 5 mg Amlodipine FDC (N=112) | 40 mg Telmisartan and 5 mg Amlodipine FDC (N=113)
Nasopharyngitis (Infections and infestations) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.